CLINICAL TRIAL: NCT01286883
Title: Prevalence of Stem Cell and Prognostic Markers in Circulating Tumor Cells of Patients With Metastatic Colorectal Cancer Undergoing Chemotherapy
Brief Title: Cancer Stem Cell Markers and Prognostic Markers in Circulating Tumor Cells
Status: Terminated | Type: Observational
Why Stopped: PI left Institution
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: PSHCI 10-066; PSHMC IRB No. 34902EP (Other: Penn State Hershey Medical Center IRB No. 34902EP)
Record Dates: First submitted 2011-01-28; First posted 2011-01-31 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2017-01

CONDITIONS: Colorectal Cancer
Keywords: stem cell markers; prognostic markers; metastatic colorectal cancer; circulating tumor cells; tumor microenvironment; colorectal cancer; advanced colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be drawn at 7 different time intervals to analyze CSC and other prognostic markers on circulating tumor cells.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Blood draws: Laboratory studies will be performed at baseline; Cycle 1, Day 1; Cycle 1, Day 7; Cycle 2, Day 1; Cycle 3, Day 1; Cycle 4, Day 1; Cycle 6, Day 1; Cycle 12, Day 1.

SUMMARY:
The study will enroll patients with metastatic colorectal cancer receiving chemotherapy. A total of approximately 22 cc of blood will be drawn during various chemotherapy infusions. Additional proposed laboratory studies may unravel important biological insights into the relationship of circulating tumor cell genomic and genetic profiles as they compare to the primary tumors. Additionally the investigators hope to gain an understanding of potential subgroups of patients that have very high numbers of circulating tumor cells or those with early relapse of circulating tumor cells after early reduction of circulating tumor cell numbers.

DETAILED DESCRIPTION:
Metastatic colorectal cancer (mCRC) has a five year survival of <10% and is the cause of death of nearly 50,000 individuals in the United States each year. Current first and second line therapies for mCRC include FOLFOX, XELOX, or FOLFIRI in combination with Bevacizumab or Cetuximab or Panitumumab, as well as Xeloda, camptosar or infusional 5-FU within various less intensive regimens for patients who cannot tolerate full-dose chemotherapy. Current practice involves evaluation of response by imaging at 2-3 months after initiation of therapy. Recent studies have demonstrated that the number of circulating tumor cells (CTCs) in the blood of patients with mCRC has independent prognostic value in terms of reflecting disease burden as well as indicating response to therapy. The use of CTC counts offers the possibility of predicting response in treated patients at an earlier time than through standard means by using CT scans. The investigators hypothesize that subsets of CTCs with cancer stem cell (CSC) markers or other known prognostic markers may improve the prognostic value of CTC evaluation in the course of therapy of patients with mCRC. The protocol will use Veridex CellSearch technology and will when possible compare this to other emerging technologies including microfluidic devices that can isolate CTCs or GFP-expressing adenoviruses that replicate in telomerase-expressing epithelial tumor cells ex-vivo. The protocol will enroll 200 patients with metastatic colorectal cancer receiving therapy. Additional proposed laboratory studies may unravel important biological insights into the relationship of CTC genomic and genetic profiles as they compare to the primary tumors. Additionally the investigators hope to gain an understanding of potential subgroups of patients that have very high numbers of CTCs or those with early relapse of CTC after early reduction of CTC numbers. The impact of this research may be in better prediction of response to mCRC therapy so that patients can be treated with second line or other experimental therapy if they are unlikely to respond to their current therapy as predicted by CTC evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of metastatic colorectal cancer, either newly diagnosed or recurrent, with measurable disease that has not been irradiated within the last 5 weeks.
* Age > 18 years old
* ECOG performance status 0-3

Exclusion Criteria:

* Patients who have received prior therapy in the last 5 weeks
* Ongoing therapy with a particular regimen that was initiated prior to enrollment and lack of availability of baseline CTC evaluation
* Patient with concurrent diagnosis of other active solid malignancies will be exclude
* Patient life expectancy of less than six weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Primary endpoint: correlation of stem cell markers on CTCs with response to therapy | 3 years
  Correlate the presence of stem cell markers and prognostic markers on circulating tumor cells with response to therapy for advanced colorectal cancer, as well as overall survival

SECONDARY OUTCOMES:
Secondary Outcome: Correlation of stem cell markers in primary tumors with stem cell markers in CTCs | 3 years
  Evaluate the primary tumor if available for stem cell markers and prognostic markers. Perform genomic analysis of CTC DNA. Compare genomic analysis of primary tumor and CTC DNA. Evaluate CTC gene expression profiles and compare with primary tumor profiles. Evaluate emerging microfluidic devices in pilot studies that use drops of blood for CTC analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Wafik S El-Deiry, MD, PhD, Principal Investigator — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
To evaluate if data is valuable

REFERENCES:
- [Background] Allen JE, El-Deiry WS. Circulating Tumor Cells and Colorectal Cancer. Curr Colorectal Cancer Rep. 2010 Oct 1;6(4):212-220. doi: 10.1007/s11888-010-0069-7. PMID 20890370